CLINICAL TRIAL: NCT00807924
Title: American Breast Laser Ablation Therapy Evaluation (ABLATE): Monitoring the Long Term Safety and Efficacy of Novilase™ Breast Interstitial Laser Therapy in Real World Application
Brief Title: American Breast Laser Ablation Therapy Evaluation
Acronym: ABLATE
Status: Completed | Type: Observational
Sponsor: Novian Health Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: BR001
Record Dates: First submitted 2008-12-11; First posted 2008-12-12 (Estimated); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Benign Breast Conditions; Breast Fibroadenomas
Keywords: Fibroadenomas; Papillomas; Breast; Minimally invasive; Interstitial laser therapy; Laser ablation; Benign; Non-cancerous; Breast lesion; Breast tumor
MeSH Terms: conditions — Fibroadenoma; Papilloma; Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this patient tracking program is to monitor long term safety and effectiveness of the Novilase™ device and method in real world application.

DETAILED DESCRIPTION:
ABLATE is a prospective, observational multi-center tracking database which will evaluate clinical outcomes from patients undergoing Novilase for benign breast conditions (i.e. fibroadenomas, papillomas, etc). Data captured will assess the potential advantages and disadvantages of the procedure as compared with lumpectomy. Tumor characteristics, equipment used, complications, patient satisfaction and cosmesis ratings will also be tracked.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis confirmed by needle core biopsy
* Tumors detected either by physical exam or imaging
* Tumors do not exceed 2 cm in diameter and measure at least 0.5 cm away from the skin and chest wall
* Single, multiple and/or bilateral tumors
* Patient has given consent prior to being treated with Novilase™

Exclusion Criteria:

* Patient is pregnant or lactating
* Hypercellularity suggestive of phyllodes
* Atypia
* Equivocal pathology report (e.g., discordance between radiographic and microscopic results)
* Fibroadenomas with stromal solidarity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing Novilase for the treatment of benign breast conditions at Novian Health affiliated breast centers.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2008-12; Primary Completion 2017-08-28 (Actual); Study Completion 2018-08-08 (Actual)

PRIMARY OUTCOMES:
To monitor and measure long term safety and effectiveness Novilase | ongoing
To help refine, improve and/or validate breast tumor best practices and standard of care | ongoing
To help establish uniform and standardized imaging, pathological assessment and ablation timing protocols | ongoing
To support the medical and patient communities through transparency--by contributing and publishing relevant, useful and meaningful data to support the development and design of future research | ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Chen, MD, Principal Investigator — Optum ProHealthcare
Locations (1):
- Columbia University Medical Center - Department of Surgery, New York, New York, United States

REFERENCES:
- [Background] Dowlatshahi K, Wadhwani S, Alvarado R, Valadez C, Dieschbourg J. Interstitial laser therapy of breast fibroadenomas with 6 and 8 year follow-up. Breast J. 2010 Jan-Feb;16(1):73-6. doi: 10.1111/j.1524-4741.2009.00830.x. Epub 2009 Oct 12. PMID 19825000
- [Background] Schwartzberg B, Lewin J, Abdelatif O, Bernard J, Bu-Ali H, Cawthorn S, Chen-Seetoo M, Feldman S, Govindarajulu S, Jones L, Juette A, Kavia S, Maganini R, Pain S, Shere M, Shriver C, Smith S, Valencia A, Whitacre E, Whitney R. Correction to: Phase 2 Open-Label Trial Investigating Percutaneous Laser Ablation for Treatment of Early-Stage Breast Cancer: MRI, Pathology, and Outcome Correlations. Ann Surg Oncol. 2018 Dec;25(Suppl 3):998. doi: 10.1245/s10434-018-6861-3. PMID 30298314
- See also: Sponsor website — http://www.novianhealth.com